CLINICAL TRIAL: NCT05132595
Title: Esketamine vs. Ketorolac for Prevention of Postoperative Pain and Cognitive Dysfunction After Total Knee Arthroplasty in Patients: a Randomized Double-blind Controlled Trial
Brief Title: Esketamine vs. Ketorolac for Prevention of Postoperative Pain and Cognitive Dysfunction After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GWang020
Record Dates: First submitted 2021-10-28; First posted 2021-11-24 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain; Postoperative Cognitive Dysfunction; Total Knee Arthroplasty
Keywords: esketamine; ketorolac
MeSH Terms: conditions — Pain, Postoperative; Postoperative Cognitive Complications | interventions — Saline Solution; Sodium Chloride; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal saline in patients (Placebo Comparator): After the induction of anesthesia, normal saline is intravenously injected in a volume of 2ml, and then a continuous infusion of 20 ml/h normal saline until starting skin suture.
  Interventions: Drug: Normal saline
- Esketamine in patients (Active Comparator): After the induction of anesthesia, esketamine is intravenously injected at 0.4mg/kg, and then a continuous infusion of 0.4mg/kg/h esketamine until starting skin suture.
  Interventions: Drug: Esketamine at high dose
- Ketorolac in patients (Active Comparator): After the induction of anesthesia, ketorolac is intravenously injected at 0.4mg/kg, and then a continuous infusion of 0.4mg/kg/h ketorolac until starting skin suture.
  Interventions: Drug: Ketorolac at high dose
- Esketamine and Ketorolac in patients (Active Comparator): After the induction of anesthesia, 0.2mg/kg esketamine and 0.2mg/kg ketorolac are intravenously injected, and then a continuous infusion of 0.2mg/kg/h esketamine and 0.2mg/kg/h ketorolac until starting skin suture.
  Interventions: Drug: Esketamine at low dose; Drug: Ketorolac at low dose

INTERVENTIONS:
Drug: Normal saline — After the induction of anesthesia, normal saline is intravenously injected in a volume of 2ml, and then a continuous infusion of 20ml/h normal saline until starting skin suture.
  Other Names: 0. 9% Sodium Chloride Injection
  Arms: Normal saline in patients
Drug: Esketamine at high dose — After the induction of anesthesia, esketamine is intravenously injected at 0.4mg/kg, and then a continuous infusion of 0.4mg/kg/h esketamine until starting skin suture.
  Other Names: Esketamine Hydrochloride Injection
  Arms: Esketamine in patients
Drug: Esketamine at low dose — After the induction of anesthesia, esketamine is intravenously injected at 0.2mg/kg, and then a continuous infusion of 0.2mg/kg/h esketamine until starting skin suture.
  Other Names: Esketamine Hydrochloride Injection
  Arms: Esketamine and Ketorolac in patients
Drug: Ketorolac at high dose — After the induction of anesthesia, Ketorolac is intravenously injected at 0.4mg/kg, and then a continuous infusion of 0.4mg/kg/h Ketorolac until starting skin suture.
  Other Names: Ketorolac Tromethamine
  Arms: Ketorolac in patients
Drug: Ketorolac at low dose — After the induction of anesthesia, Ketorolac is intravenously injected at 0.2mg/kg, and then a continuous infusion of 0.2mg/kg/h Ketorolac until starting skin suture.
  Other Names: Ketorolac Tromethamine
  Arms: Esketamine and Ketorolac in patients

SUMMARY:
Purpose:

To compare esketamine and ketorolac separately and in combination to prevent postoperative pain and cognitive dysfunction after total knee arthroplasty

DETAILED DESCRIPTION:
With the increase in human life span, orthopedic injuries and subsequent repair surgery have become a major health problem which impairs the life quality of patients and burdens healthcare systems worldwide. Poor post-surgical pain control is a leading factor that hinders the physical rehabilitation and musculoskeletal functional recovery, and causes acute cognitive impairment and chronic pain syndrome. Therefore, prophylaxis of postoperative pain is indispensable to postoperative comfort and satisfaction. There is no denying the fact that pathologic pain is related to central glutaminergic system and N-methyl-d-aspartate (NMDA) receptor activation induced central sensitization. Also, it is previously reported that neuroinflammation is associated with pain development and cognitive dysfunction. Ketamine, a NMDA receptor antagonist, is effective in reversing NMDA receptor activation underlying pain states. But the side effects of ketamine limit its clinical application, such as gibberish and agitation. It is clarified that esketamine has lower side effects than ketamine and that antinociception of esketamine is stronger than ketamine. The following study is carried out to evaluate whether esketamine and ketorolac can prevent postoperative pain and cognitive impairment after total knee arthroplasty in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo total knee arthroplasty under a short general anesthesia of less than 2 hours
2. Subject's American Society of Anesthesiologists physical status is I-II.
3. The subject's parent/legally authorized guardian has given written informed consent to participate.

Exclusion Criteria:

1. Subject has a diagnosis of bronchial asthma, coronary heart disease, severe hypertension, renal failure or liver failure.
2. Subject has a diagnosis of Insulin dependent diabetes.
3. Subject is allergy and contraindication to esketamine or ketorolac.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre- existing therapy with opioids.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Subject is pregnant or breast-feeding.
7. Subject is obese (body mass index >30kg/m^2).
8. Subject is incapacity to comprehend pain assessment and cognitive assessment.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid Consumption | 72 hours after surgery
  Each patient was administered analgesics using a PCA (Patient-controlled analgesia) pump containing sufentanil in normal saline after leaving PACU (Postanesthesia care unit). Sufentanyl cumulative consumption is recorded 72 hours postoperatively

SECONDARY OUTCOMES:
Pain Score (NRS) after movement | 72 hours after surgery
  The pain score after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
Time of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Total Dose of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Mini-Mental State Examination (MMSE) | 72 hours after surgery
  Cognitive performance was assessed with 0-30 points Mini-Mental State Examination (MMSE) scale. Greater scores means better outcome.
The incidence of Side Effects | 72 hours after surgery
  The number of patients with post-operative side effects including nausea, vomiting, dizziness, headache, shivering, and pruritus was recorded 72 hours after surgery.
The levels of TNF-a in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of cytokine TNF-a using ELISA kits.
The levels of chemokine CXCL1 in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of chemokine CXCL1 using ELISA kits.
The levels of neuron specific enolase (NSE) in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of neuron specific enolase (NSE) using electrochemilumiscence kit.
The levels of S-100 calcium-binding protein B in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of S-100 calcium-binding protein B using electrochemilumiscence kit.
The levels of cortisol in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of cortisol using electrochemilumiscence kit.
Pain Score (NRS) at rest | 72 hours after surgery
  The pain score at rest was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
The levels of chemokine CCL7 in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of chemokine CCL7 using ELISA kits.
The levels of IL-18 in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of cytokine IL-18 using ELISA kits.
The levels of IL-23 in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of cytokine IL-23 using ELISA kits.
The levels of IL-17 in blood | 72 hours after surgery
  Blood samples are collected to measure the levels of cytokine IL-17 using ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No